CLINICAL TRIAL: NCT02956200
Title: A Randomised Controlled Trial of Combinating an Immune Modulator Fingolimod With Alteplase Bridging With Mechanical Thrombectomy in Acute Ischemic Stroke
Brief Title: Combinating Fingolimod With Alteplase Bridging With Mechanical Thrombectomy in Acute Ischemic Stroke
Acronym: FAMTAIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shaoxing People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huzhou Center Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Jinhua Center Hospital (Unknown); Taizhou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YAN-2016-047
Record Dates: First submitted 2016-10-11; First posted 2016-11-07 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2016-09

CONDITIONS: Stroke; Inflammation
Keywords: Fingolimod Hydrochloride; Intravenous thrombolysis; Mechanical thrombectomy; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Inflammation; Ischemic Stroke | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fingolimod with standard therapy (Experimental): Patients will be treated with standard alteplase bridging and mechanical thrombectomy with fingolimod.
  Interventions: Drug: Fingolimod
- standard therapy (No Intervention): Patients will be treated with standard alteplase bridging and mechanical thrombectomy.

INTERVENTIONS:
Drug: Fingolimod — Patients randomized to fingolimod will also receive oral fingolimod (Gilenya, Novartis) at a dosage of 0.5 mg once daily, for three consecutive days, with the first dose being given at the time in which patients are enrolled which is about one hour prior to mechanical thrombectomy.
  Other Names: Fingolimod Hydrochloride
  Arms: fingolimod with standard therapy

SUMMARY:
Proof-of concept clinical trials have indicated that the sphingosine-1-phosphate receptor modulator fingolimod may be efficacious in attenuating brain inflammation and improving clinical outcomes in patients with AIS as a single therapy beyond 4.5 hours of disease onset, or in combination with alteplase within 4.5 hours of disease onset. So in this study the investigators try to determine whether the addition of fingolimod, administered within 6 hours after the onset of symptoms in patients receiving alteplase bridging with mechanical thrombectomy, improves radiologic and clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, blinded endpoint (PROBE) design clinical trial, in multiple stroke centers of China. The total sample size will be 98. Patients being treated with standard alteplase bridging and mechanical thrombectomy will be randomly assigned in a 1:1 ratio to receive oral fingolimod or standard care. The primary outcome will be the salvaged ischemic tissue from baseline to day 7. AIS patients with proximal cerebral arterial occlusions will have CT perfusion (CTP) before treatment, and multimodal MRI including diffusion and MR perfusion (MRP) at 24 hours and 7 days after receiving treatment. Clinical outcomes will be assessed using the National Institutes of Health Stroke Scale score (NIHSS) at baseline, day 1 and day 7 and the modified Rankin Scale (mRS) at 90 days. Circulating lymphocyte counts will be monitored with FACS at baseline, day 1 and day 7 to confirm the biological activity of fingolimod.

Patients aged between 18 and 85 with anterior circulation AIS who are eligible for alteplase and mechanical thrombectomy commenced within 6 hours of stroke onset will be enrolled if they present with an infarct core volume between 15-100 mL with at least 20% mismatch (as evaluated by CTP) and intracranial occlusion in proximal cerebral arteries. Exclusion criteria are (1) standard contraindications to alteplase or mechanical thrombectomy; (2) evidence of other diseases of the CNS; (3) pre-existing neurologic disability (a score greater than 2 on the mRS); (4) swallowing difficulties that would prevent administration of oral fingolimod; (5) patients with any history of bradyarrhythmia, atrioventricular block or current use of beta-blockers or verapamil; (6) concomitant use of antineoplastic, immunosuppressive or immune modulating therapies; (7) macular edema.

As standard care, all patients will receive standard dose intravenous alteplase (0.9 mg per kilogram, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg) and mechanical thrombectomy delivered at the site of intracranial vessel occlusion. Patients randomized to fingolimod will also receive oral fingolimod (Gilenya, Novartis) at a dosage of 0.5 mg once daily, for three consecutive days, with the first dose being given at the time in which patients are enrolled which is about one hour prior to mechanical thrombectomy.

The kinetics of lymphocyte subset alteration will be monitored in whole-blood samples from all fingolimod- treated patients at the baseline, which will precede the first dose, day 1 and day 7. Mononuclear cells will be isolated from the whole-blood specimens and stained with antibodies to CD4-FITC, CD8-PE, CD19-PerCP, CD56-PE (BD Biosciences, Franklin Lakes, NJ, USA). Data will be acquired using a FACS Caliber (Becton Dickinson Immunocytometry Systems, San Jose, CA, USA) and analyzed with Flow Jo software (Tree Star, Ashland, OR, USA).

The primary outcome is salvaged ischemic tissue((baseline ischemic lesion - 7d infarction lesion)/ baseline ischemic lesion) from baseline to day 7. Secondary outcomes are the growth in infarct volume between 24 hour DWI and day 7 FLAIR imaging, the penumbral salvage volume (baseline hypoperfusion volume - 24-hours infarct volume) between the baseline and day 1, the frequency of parenchymal hemorrhage (PH) at day 1 and the extent of clinical improvement at day 1 as measured by the change on the NIHSS score from baseline to day 1, the extent of clinical improvement from day 1 to day 7. The tertiary outcomes are the probability of excellent recovery at day 90 (mRS 0-1), independent recovery (mRS 0-2) and ordinal analysis of the modified Rankin scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with anterior circulation acute ischaemic stroke who are eligible for alteplase and mechanical thrombectomy commenced within 6 hours of stroke onset.
2. Patient, family member or legally responsible person depending on local ethics requirements has given informed consent.
3. Patient"s age is 18-85 years.
4. Arterial occlusion on CTA of the ICA, M1 or M2.
5. Imaging inclusion criteria: infarct core volume between 15-100 mL with at least 20% mismatch (as evaluated by CTP).

Exclusion Criteria:

1. Standard contraindications to alteplase or mechanical thrombectomy.
2. Evidence of other diseases of the CNS.
3. Pre-existing neurologic disability (a score greater than 2 on the mRS).
4. Swallowing difficulties that would prevent administration of oral fingolimod.
5. Patients with any history of bradyarrhythmia, atrioventricular block or current use of beta-blockers or verapamil.
6. Patients with serious acute or chronic infection, or hepatic injury (over 3 times value of normal ALS or AST).
7. Concomitant use of antineoplastic, immunosuppressive or immune modulating therapies.
8. Macular edema.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
salvaged ischemic tissue index (%) | from baseline to 7 day
  100*(baseline CTP ischemic lesion (mL) - 7 day DWI infarction lesion (mL))/ baseline CTP ischemic lesion (mL)

SECONDARY OUTCOMES:
the growth in infarct volume (mL) | from 24 hour to 7 day
  24 hour DWI infarct volume (mL) - 7 day FLAIR infarct volume (mL)
the penumbral salvage volume (mL) | from baseline to 1 day
  (baseline CTP hypoperfusion volume (mL) - 24 hour DWI infarct volume (mL))
the frequency of parenchymal hemorrhage (PH) (%) | at day 1
  the presence of PH is defined according the standard from ECASS-2 study
the change on the NIHSS score | from baseline to 1 day
  baseline NIHSS score - 1 day NIHSS score
the change on the NIHSS score | from baseline to 7 day
  baseline NIHSS score - 7 day NIHSS score
excellent recovery | at day 90
  modefied Rankin Scale (mRS) score of 0-1
independent recovery | at day 90
  mRS score of 0-2

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, MD,PhD, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided